CLINICAL TRIAL: NCT04798937
Title: A RCT Using Motivational Interviewing to Improve Self Management in Youth With Type 1 Diabetes
Brief Title: Motivational Interviewing to Improve Self Management in Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sousse (Other)
Responsible Party: Principal Investigator, Kawther Al ksir, Principal Investigator, Université de Sousse
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 140221
Record Dates: First submitted 2021-03-07; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: type1diabetes
Keywords: adolescent; transition to adult care; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: 78 were screened and 66 youth were randomized to 2 groups of 33 each and followed for 6 months with data collection at time zero, 3 months and 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Youth in this group received usual care, consisting of medical consultations, in combination with a health education program based on motivational interviewing provided by a nurse
  Interventions: Other: Motivational interviewing
- Control group (No Intervention): Youth in this group received usual care only consisting of medical consultations

INTERVENTIONS:
Other: Motivational interviewing — a health education program based on motivational interviewing provided by a nurse
  Arms: Intervention group

SUMMARY:
A brief, nurse-led educational intervention using motivational interviewing substantially improved general and disease-specific self-management skills in youth with type 1 diabetes.

DETAILED DESCRIPTION:
Introduction and Objectives: For youth with chronic health conditions, adolescence is associated with a deterioration of disease self-management and poor health outcomes. Effective interventions are needed to prepare youth for transition to adulthood and adult care. To prospectively assess the impact of an education program based on motivational interviewing on self-management skills and glycemic control in youth with Type 1 diabetes (T1D).

Methods: After parental consent and youth assent, investigators prospectively randomized 66 adolescents 13-18 years old with type 1 diabetes to either usual care (regular medical consultation) or usual care supplemented by sessions with a nurse educator using a motivational interviewing (MI) approach and goal setting based on responses to the Transition Readiness Assessment Questionnaire (TRAQ) and T1D specific self-management skills. Primary outcomes were TRAQ change scores and HbA1c levels between baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with type 1 diabetes
* Having an age between 13 and 18 years

Exclusion Criteria:

* Having a neurological disability (epilepsy, autism)
* Having a significant intellectual delay, which might have affected their ability to understand the content of the program

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Transition Readiness Assessment Questionnaire (TRAQ) scores | Change from Baseline TRAQ score at 6 months
  The TRAQ includes 20 items divided into five subscales: 1) Appointment keeping (7 questions; e.g., Do you call the doctor's office to make an appointment?) 2) Tracking health issues (4 questions; e.g., Do you keep a calendar or list of medical and other appointments?); 3) Managing medications (4 questions; e.g., Do you know what to do if you are having a bad reaction to your medications?); 4) Talking with healthcare providers (2 questions; e.g. Do you tell the doctor or nurse what you are feeling?); 5) Managing daily activities (3 questions; e.g. Do you help plan or prepare meals/food?). Each question has the same Liker response set from 1 to 5 using the Stages of Change Transtheoretical Model as a framework. A minimum score of ''1'' is assigned to the responses 'No, I don't know how' while a maximum score of '' 5 '' is assigned to responses labeled "Yes, I always do it when I need it." Higher scores mean better outcome.

SECONDARY OUTCOMES:
Hemoglobin glycated values | Change from Baseline Hemoglobin glycated values at 6 months
  Hemoglobin glycated values

CONTACTS AND LOCATIONS:
Overall Officials: David Wood, Dr, Study Director — East Tennessee State University
Locations (1):
- Farhat Hached University Hospital, Sousse, Tunisia

REFERENCES:
- [Derived] Al Ksir K, Wood DL, Hasni Y, Sahli J, Quinn M, Ghardallou M. Motivational interviewing to improve self-management in youth with type 1 diabetes: A randomized clinical trial. J Pediatr Nurs. 2022 Sep-Oct;66:e116-e121. doi: 10.1016/j.pedn.2022.05.001. Epub 2022 May 12. PMID 35568602